CLINICAL TRIAL: NCT00266123
Title: A Randomized Open-Label Study to Compare the Safety and Efficacy of Two Different Sirolimus Regimens With a Tacrolimus + Mycophenolate Mofetil Regimen in De Novo Renal Allograft Recipients
Brief Title: Study Comparing Two Sirolimus Regimens vs. Tacrolimus and Mycophenolate Mofetil Regimen in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-101497
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Graft Rejection; Kidney Failure; Kidney Transplant
Keywords: Kidney Failure; Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
To demonstrate the superiority of SRL + TAC elimination + corticosteroids (Group I) and SRL + MMF + corticosteroids (Group II) to TAC + MMF + corticosteroids (Group III) with respect to renal allograft function at month 12 post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* End-stage renal disease with subjects scheduled to receive a primary or secondary renal allograft from a cadaveric donor, from a living-unrelated mismatched donor, or from a living-related mismatched donor. Unreported HLA values will be considered a match.
* Women of childbearing potential must have a negative serum pregnancy test before administration of assigned treatment and agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months following discontinuation of assigned treatment.

Other inclusions apply.

Exclusion Criteria:

* Evidence of active systemic or localized major infection.
* Known hypersensitivity to SRL or its derivatives, macrolide antibiotics, corticosteroids, TAC or MMF.
* Multiple organ transplants (i.e., prior or concurrent transplantation of any organs other than renal transplant).

Other exclusions apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2004-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Kidney function at 52 weeks after transplantation.

SECONDARY OUTCOMES:
Kidney function at 26, 78 and 104 weeks after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth Reseach; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com; Trial Manager, Principal Investigator — For United Kingdom, ukmedinfo@wyeth.com